CLINICAL TRIAL: NCT00145808
Title: Prospective Controlled Assessment of Wireless Capsule Endoscopy (WCE) in Ulcerative Colitis (UC)
Brief Title: Wireless Capsule Endoscopy in Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Prometheus Laboratories (Industry); American College of Gastroenterology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 13215A
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative

INTERVENTIONS:
Device: Given® Diagnostic System

SUMMARY:
Based on the inaccuracies of the current classification scheme for inflammatory bowel disease (IBD), the failure of surgical pouches and the findings of retrospective observational trials to date, we hypothesize that a significant proportion of patients with UC will have small bowel involvement that will result in a change in diagnosis to CD or the recognition of a new phenotype of IBD. The aim of this study is to determine the prevalence of small bowel pathology in patients diagnosed with UC using WCE. This information will aid in the current efforts to re-classify IBD using improved endoscopic and imaging technologies, genetic information and serologic information.

DETAILED DESCRIPTION:
Subjects will undergo both a blood draw and a wireless capsule endoscopy (WCE).

The blood draw will occur in the GI procedure unit on the day of subjects exam.

WCE: Subject will only consume a clear liquid diet after noon the day prior to the exam. No food or beverage consumption any after 10 PM on the day before examination. Not oral medications after 12 AMon the day of exam (8 hours before subject's exam).

Day of exam, subject will report to the endoscopy unit. At that time, subject will be prepared for examination by doctor who will apply a sensor array to the abdomen with adhesive sleeves. In addition, a waist belt device that holds the data recorder will be fitted to subject. Subjects will swallow the capsule endoscope. The capsule endoscope passes naturally through digestive tract while transmitting video images to the data recorder worn on the belt for approximately eight hours. At this point, subjects will be free to leave the University of Chicago hospital until they return eight hours later for disconnection of the recording equipment.

Two hours after ingestion of the capsule, subject will be able to resume a clear liquid diet. Four hours after the study's start time, subject will be able to resume a regular diet ( solid foods). At this time, subject will also be able to resume taking oral medications.

After eight hours, subject will return to the endoscopy suite (DCAM 6H) for disconnection of the recording equipment (sensor array, data recorder, and belt). The time that the capsule was ingested, eating and drinking times, and disconnection time as well as any discomfort subject experienced will be recorded.

Subject will be contacted 72 hours after the examination to confirm passage of the capsule. If they have not reported passage of the capsule with this time, subject will undergo an abdominal radiograph in order to determine whether or not the capsule has passed.

Subjects will be asked to identify a non-relative control (spouses are acceptable) within five years of their age and of similar background without Ulcerative Colitis. There is an Information Handout that participating subjects will give to friends interested in participating. If the subject does not find anyone, they may still participate in this research study. The study staff will try to find someone for them.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the "disease" arm include a clinical impression of ulcerative colitis that includes assessment of the colon by colonoscopy and biopsy and assessment of the terminal ileum either by ileoscopy or by small bowel radiograph or enteroclysis. Subjects in the "control" arm will only be included if they do not carry the diagnosis of UC or CD, have not had previous gastric or small bowel surgery and are free of gastrointestinal symptoms including unexplained abdominal pain, diarrhea or gastrointestinal bleeding.

Exclusion Criteria:

A known bowel obstruction, fistula or stricture, a permanent pacemaker and/or implantable defibrillator, history of a swallowing disorder, inability to provide informed consent, pregnancy, the use of aspirin or non-steroidal anti-inflammatory drugs (NSAIDs) within the past 30 days, known celiac disease, known terminal ileal disease on ileoscopy and a history of occult or obscure gastrointestinal bleeding of unclear etiology. In menstruating females, a urine HCG will be performed on the day they arrive for the study (prior to ingestion of the capsule), if fourteen (14) days or more have elapsed since their last menstrual period. If subject reports they are menopausal, a urine HCG will be performed unless subject has had no menses during the past two years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2005-06; Primary Completion 2007-06 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Assess the prevalence of small bowel abnormalities in UC patients compared to controls.

SECONDARY OUTCOMES:
Ensure safety of subjects by confirming passage of the capsule.

CONTACTS AND LOCATIONS:
Overall Officials: David Rubin, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States